CLINICAL TRIAL: NCT04108949
Title: Tuning in to Kids: an Effectiveness Evaluation of Emotion Coaching to Parents and Daycare Teachers of At-risk Young Children
Brief Title: Small Children, Big Emotions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to consequences of the Covid-19 pandemic, which made it impossible to complete the trial in a timely manner and in accordance with the study protocol
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other); University of Melbourne (Other); Extrastiftelsen (Other)
Responsible Party: Principal Investigator, Marianne Aalberg, Researcher, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/02391
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Emotional Disturbances
MeSH Terms: conditions — Affective Symptoms | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with two arms.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to treatment condition and receive no information about which treatment the participant will receive or have received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tuning in to Kids (Experimental): Eight weekly two-hour sessions delivered in groups of up to six parents.
  Interventions: Behavioral: Tuning in to Kids
- Treatment as usual (Active Comparator): Treatment as usual, may consist of any psychosocial intervention the therapist sees fit, which is the type of intervention the participants ordinarily receives in the participating clinics. No limit on number of sessions or format of delivery.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Tuning in to Kids — A psychosocial intervention focusing on emotion socialization and emotion coaching.
  Arms: Tuning in to Kids
Behavioral: Treatment as usual — See description included in arm/Group description.
  Arms: Treatment as usual

SUMMARY:
The study is a randomized controlled trial evaluating the clinical and cost-effectiveness of Tuning in to Kids (TIK) compared to treatment as usual (TAU). Participants are recruited among referred children aged 2-5 years with difficulties with emotion regulation. The study setting is Child and Adolescent Mental Health Services clinics. Parents of children randomized to TIK will attend 8 two-hourly group sessions. A brief version of TIK will be offered to the child's daycare teacher. Participants are assessed at baseline, week 12 and month 9 after inclusion. The primary clinical outcome is Coping with Toddlers' Negative Emotions Scale.

ELIGIBILITY:
Inclusion Criteria:

* Referred children aged 2-5 years
* The child is enrolled in daycare
* The child is displaying problems with emotional dysregulation

Exclusion Criteria:

* Parent not sufficiently proficient in Norwegian Language to Complete assessment
* Child Protective Services have ongoing assessment where the outcome may be that the child will be placed in care outside of the home of the biological parent(s) or other current caregiver
* The child has already been diagnosed with an autism spectrum disorder

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Coping with Toddlers' Negative Emotion Scale | CTNES will be completed at baseline, post treatment (week 12) and follow-up month 9 after inclusion) to evaluate change from baseline to post-treatment and follow-up.
  A measure of parental behaviors in respond to toddlers' emotions. CTNES consists of 12 hypothetical situation where parents rate their likelihood of responding in six different ways on a scale from 1 (very unlikely) to 7 (very likely).

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Aalberg, PhD, Principal Investigator — University Hospital, Akershus
Locations (3):
- Norway (3):
  - BUP Øvre Romerike, Jessheim
  - BUP Grorud, Oslo
  - Nic Waals Institutt, Oslo